CLINICAL TRIAL: NCT07274371
Title: Effects of Brahmi-Gotu Kola Oil Padabhyanga (Foot Massage) on Sleep and Mood Disturbances in Perimenopausal Women: a Pragmatic, Single-blind, Pilot Randomized Controlled Comparative Trial
Brief Title: A Study Comparing the Effects of Two Types of Natural Oils Used in a Bedtime Foot Massage Routine on Sleep and Emotional Well-Being in Perimenopausal Women.
Acronym: BG-SLEEP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saipriya Gowrishankar (Other)
Collaborators: Maharishi International University (Other)
Responsible Party: Sponsor-Investigator, Saipriya Gowrishankar, Principal Investigator and PhD Candidate in Physiology, Maharishi International University
Organization: Maharishi International University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BRAHMI-GOTUKOLA OIL- RCT-01
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Sleep Disturbances in Perimenopause
Keywords: perimenopause; sleep disturbance
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Intervention Model Description: This pragmatic randomized trial evaluates the effects of a nightly 10-minute self-administered Pada Abhyanga (foot massage) routine among perimenopausal women. All participants perform the same massage protocol, and are randomly assigned to use either Brahmi- Gotukola oil or plain sesame oil. The delivery, frequency, and duration of the intervention are identical in both groups; only the oil differs. Participants remain in their assigned group for the full study period, with no crossover.
Who Masked: Participant
Masking Description: It is a single blinded trial so the participants does not know which noil they are using.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brahmi-Gotukola oil Padabhyanga( foot massage) (Experimental): Participants apply Brahmi-Gotukola oil to both feet and perform a 10-minute Ayurvedic foot massage (Pada Abhyanga) once daily at bedtime for 14 consecutive days. Approximately 1 teaspoon (5 mi) of warm oil is applied to each foot. Massage is performed for 5 minutes per foot with focused strokes on the center of the foot, base of the big toe and other toes, web spaces, medial and lateral borders, ankle joint, Achilles tendon, and the dorsum. After massage, excess oil may be wiped with a paper towel to reduce slipperiness, and cotton socks may be worn.
  Interventions: Behavioral: Brahmi-Gotukola oil padabhyanga
- Sesame oil padabhyanga ( foot massage) (Active Comparator): Participants apply sesame oil to both feet and perform the same 10 minute Ayurvedic foot massage (Padabhyanga) once daily at bedtime for 14 consecutive days. Approximately 1 teaspoon (5 ml) of oil is applied to each foot. The identical 5 minute per foot massage protocol is followed with emphasis on the center of the foot, toe bases, web spaces, medial/lateral borders, ankle joint, Achilles tendon, and dorsum. After massage, excess oil may be wiped with a paper towel, and cotton socks may be worn to prevent slipping.
  Interventions: Behavioral: Sesame oil Padabhyanga

INTERVENTIONS:
Behavioral: Brahmi-Gotukola oil padabhyanga — The intervention consists of applying Brahmi-Gotukola oil to both feet followed by a 10-minute Ayurvedic foot massage (Padabhyanga), performed once daily at bedtime for 14 consecutive days. Approximately 1 teaspoon (5 ml) of oil is applied to each foot. Massage is performed for 5 minutes per foot, focusing on the center of the foot, the base of the big toe and other toes, the web spaces, medial and lateral borders, the ankle joint, Achilles tendon, and the dorsum of the foot. After massage, excess oil may be gently wiped with a paper towel to reduce slipperiness, and participants may optionally wear cotton socks to prevent slipping. Massage is done about 20-30 minute before bed time , sitting in a quiet place. Intervention done after washing both feet. A parallel comparison group performs the same procedure using sesame oil instead of Brahmi-Gotu Kola oil.
  Arms: Brahmi-Gotukola oil Padabhyanga( foot massage)
Behavioral: Sesame oil Padabhyanga — Participants apply sesame oil to both feet and perform the same 10-minute Ayurvedic foot massage (Padabhyanga) once daily at bedtime for 14 consecutive days. Approximately 1 teaspoon (5 ml) of oil is applied to each foot. The identical 5-minute per foot massage protocol is followed with emphasis on the center of the foot, toe bases, web spaces, medial/lateral borders, ankle joint, Achilles tendon, and dorsum. After massage, excess oil may be wiped with a paper towel, and cotton socks may be worn to prevent slipping.
  Arms: Sesame oil padabhyanga ( foot massage)

SUMMARY:
This study is being done to find out whether a nightly 5-minute foot massage (Padabhyanga) using Brahmi-Gotukola oil can help women ages 40 to 55 sleep better and feel calmer during perimenopause. Perimenopause is the time when periods start to change and many women begin to experience sleep problems and mood changes. The study will also compare Brahmi-Gotukola oil to organic sesame oil, which will be used as the control oil.

Participants will do a simple guided 10-minute foot massage at home every night for 2 weeks using either Brahmi-Gotukola oil or organic sesame oil. They will fill out a short sleep log each morning to track their sleep. Before starting the study and again at the end of the 2-week period, they will complete questionnaires about their sleep and mood. Additional follow-up questionnaires will be completed in the 3rd and 4th weeks to see if any improvements continue even after the massage period is over.

This study aims to:

See whether Brahmi-Gotukola oil foot massage improves sleep in women experiencing perimenopausal sleep problems.

Find out whether Brahmi-Gotukola oil foot massage helps with mood and emotional well-being.

Compare Brahmi-Gotukola oil foot massage with sesame oil foot massage to determine whether Brahmi oil provides more benefits for sleep and mood.

DETAILED DESCRIPTION:
Sleep disturbances and mood changes are commonly reported during the perimenopausal transition due to fluctuating ovarian hormones, alterations in circadian rhythm, and increased vulnerability to psychological stress. Many women prefer non-pharmacological interventions for sleep support, particularly those that can be performed at home, are low-risk, and do not interfere with daily responsibilities. Ayurveda describes Padabhyanga (foot massage) as a calming practice traditionally used to improve sleep , stabilize the nervous system, and support mental well-being. Brahmi (Bacopa monnieri) and Gotu Kola (Centella asiatica) are herbs used in classical Ayurvedic formulations and are known for their calming, sleep promoting actions. However, there is limited clinical research evaluating their effects on sleep and mood specifically in oil form especially in perimenopausal women.

This randomized controlled trial will evaluate whether a nightly 5-minute Padabhyanga using Brahmi-Gotu Kola oil can improve sleep quality and mood disturbances in women aged 40-55 experiencing perimenopausal changes. The trial will compare Brahmi-Gotukola oil to organic sesame oil, which is used as the control due to its neutral and widely accepted Ayurvedic use without the specific medhya (mind-supportive) actions attributed to Brahmi. The intervention will be self-administered at home for 14 consecutive nights.

Participants will complete baseline questionnaires assessing sleep quality and mood before the intervention begins. A short daily sleep log will be completed each morning during the 2-week intervention period to track changes in subjective sleep experience. Outcome assessment will be repeated immediately after the 2-week intervention, followed by two additional follow-up questionnaires in the 3rd and 4th weeks. The purpose of the follow-up assessments is to measure whether any observed improvements persist beyond the intervention period.

This study will generate preliminary evidence on the effectiveness of Ayurvedic Padabhyanga with Brahmi-Gotukola oil as a low-risk, self-care nighttime practice for perimenopausal women. Findings may support future larger-scale trials and may provide a practical, culturally relevant, and accessible approach to improving sleep quality and emotional well-being without pharmaceutical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 40 to 55 years.
* Perimenopausal stage according to Stages of reproductive aging workshop +10 with menstrual irregularity PSQI scores above 5.
* Ability to understand and respond to study questions in English
* Willingness to participate in the study

Exclusion Criteria:

* Participants attained menopause.
* Current use of Hormone Replacement Therapy
* Current Psychiatric disorders like bipolar disorder and other severe mental illness that may interfere with partici[pation.
* Use of any anxiolytics, antidepressants
* History of Oopherectomy or hysterectomy .
* Conditions limiting foot massage include active foot injury, severe varicose vein, oprn wounds or any skin infection on the feet
* Any known allergy to sesame seeds
* Any other serious medical conditions according to investigators judgement that would ,make participation unsafe.

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Eligibility for this study is limited to individuals who are biologically female and experiencing the perimenopausal transition showing irregularities in their monthly periods. Because the study investigates physiological changes that occur only in biological females during perimenopause, participants must have been assigned female at birth. Individuals who identify as women but were not assigned female at birth, as well as individuals who were assigned female at birth but do not experience menstrual physiology, are not eligible.
Enrollment: 30 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in PSQI score from baseline to day 14 | Baseline to 14 days after intervention
  The Pittsburgh Sleep Quality Index (PSQI) will be administered at baseline (prior to intervention) and after 14 days of daily foot massage. This is a validated questionnaire that assesses sleep quality over the previous 1-month period, here adapted to a 2-week study duration. It includes 19 self-rated items generating a global score from 0 to 21, with higher scores indicating poorer sleep quality. A global score of 5 or more indicates clinically significant sleep disturbance. Change in total Pittsburg sleep quality index score will be calculated by subtracting Pretest score from Post test score.
Improvement in PSQI score from baseline to post test | Baseline ( preintervention) and 14 days after starting the intervention
  The Pittsburgh Sleep Quality Index (PSQI) will be administered at baseline (prior to intervention) and after 14 days of daily foot massage. The PSQI is a validated questionnaire that assesses sleep quality over the previous 1-month period, here adapted to a 2-week study duration. It includes 19 self-rated items generating a global score from 0 to 21, with higher scores indicating poorer sleep quality. A global PSQI score >5 indicates clinically significant sleep disturbance. Change in total PSQI score will be calculated by subtracting post-intervention score from baseline score.

CONTACTS AND LOCATIONS:
Overall Officials: Saipriya Gowrishankar, Principal Investigator — Maharishi International University
Locations (1):
- Maharishi International University, Fairfield, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data will not be made publicly available. Data will be analyzed and reported only in aggregate form for scientific publications and presentations. No individual-level datasets will be shared outside of the research team due to institutional data privacy policies and participant consent limitations.

REFERENCES:
- [Background] Sarhyal A, Chate S, Tubaki BR, Thakur R. Efficacy of Brahmi vati and Aswagandharista in major depressive disorder: A randomized controlled trial. J Ayurveda Integr Med. 2024 Nov-Dec;15(6):101022. doi: 10.1016/j.jaim.2024.101022. Epub 2024 Dec 3. PMID 39631219
- [Background] Kravitz HM, Janssen I, Bromberger JT, Matthews KA, Hall MH, Ruppert K, Joffe H. Sleep Trajectories Before and After the Final Menstrual Period in The Study of Women's Health Across the Nation (SWAN). Curr Sleep Med Rep. 2017 Sep;3(3):235-250. doi: 10.1007/s40675-017-0084-1. Epub 2017 Aug 5. PMID 28944165